CLINICAL TRIAL: NCT00420342
Title: A Double Blind, Randomized, Active-control Study to Evaluate Effects of Drospirenone/Estradiol (Angeliq) and Medroxyprogesterone Acetate/Conjugated Equine Estrogen (Prempro) on Blood Pressure and Sodium Sensitivity in Postmenopausal Women With Prehypertension
Brief Title: Effects of Angeliq and Prempro on Blood Pressure and Sodium Sensitivity in Postmenopausal Women With Prehypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 91507; 310522 (Other: Company internal)
Record Dates: First submitted 2007-01-09; First posted 2007-01-11 (Estimated); Results first posted 2010-01-20 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Postmenopause; Hypertension; Pre-Hypertension
Keywords: Pre-Hypertension in Postmenopausal Women
MeSH Terms: conditions — Hypertension; Prehypertension | interventions — estradiol-drospirenone combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 0.5mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) (Experimental): 0.5 mg drospirenone/1.0 mg 17β-estradiol for 8 weeks (8 weeks plus 3 days for sodium sensitivity subjects)
  Interventions: Drug: Drospirenone/17ß-estradiol (Angeliq, BAY86-4891)
- 2.0mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) (Experimental): 2.0 mg drospirenone/1.0 mg 17β-estradiol for 8 weeks (8 weeks plus 3 days for sodium sensitivity subjects)
  Interventions: Drug: Drospirenone/17ß-estradiol (Angeliq, BAY86-4891)
- 1.5 mg MPA / 0.3 mg CEE (Prempro) (Active Comparator): 1.5 mg medroxyprogesterone acetate/0.3 mg conjugated equine estrogen for 8 weeks (8 weeks plus 3 days for sodium sensitivity subjects)
  Interventions: Drug: SH K 00641 C - Medroxyprogesterone acetate / conjugated equine (Prempro TM)

INTERVENTIONS:
Drug: Drospirenone/17ß-estradiol (Angeliq, BAY86-4891) — SH K 00641 A -Active study medication encapsulated tablet
  Arms: 0.5mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891)
Drug: Drospirenone/17ß-estradiol (Angeliq, BAY86-4891) — SH K 00641 B - Active study medication encapsulated tablet
  Arms: 2.0mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891)
Drug: SH K 00641 C - Medroxyprogesterone acetate / conjugated equine (Prempro TM) — Active control encapsulated tablet
  Arms: 1.5 mg MPA / 0.3 mg CEE (Prempro)

SUMMARY:
The main purpose of this study is to compare the effects of treatment of two different formulations of Angeliq® and Prempro on blood pressure in post-menopausal women with prehypertension.

DETAILED DESCRIPTION:
This study has previously been posted by Berlex, Inc. Berlex, Inc. has been renamed to Bayer HealthCare Pharmaceuticals, Inc.Bayer HealthCare Pharmaceuticals, Inc. is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

- Postmenopausal women 45 - 65 years old with prehypertension

Exclusion Criteria:

- Hormone therapy (estrogen/progestin)

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2007-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (9):
- United States (9):
  - Greenbrae, California
  - San Diego, California
  - Daytona Beach, Florida
  - Miami, Florida
  - Paw Paw, Michigan
  - Las Vegas, Nevada
  - Philadelphia, Pennsylvania
  - Columbia, South Carolina
  - Arlington, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject enrollment began on 16-Jan-2007 and lasted over a period of 6 months at 10 study centers in the U.S. There was no enrollment at 2 sites (108 and 110). Site 102 enrolled 14 subjects and site 105 enrolled 56 subjects (28 of whom consented to the sodium sensitivity analysis). All other sites enrolled 7 or fewer subjects.
Pre-assignment Details: Screening involved office cuff BP measurements at 3 visits to evaluate prehypertension. Of the 178 enrolled, 86 subjects were screen failures. The full analysis and safety sets had 90 subjects who took at least 1 dose of study medication (2 subjects did not confirm if they ever took the study medication).
Period: Overall Study
Arm/Group | 0.5mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) | 2.0mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) | 1.5 mg MPA / 0.3 mg CEE (Prempro)
Started | 30 | 33 | 29
Received Treatment | 29 (1 subject did not confirm if she ever took the study medication.) | 32 (1 subject did not confirm if she ever took the study medication.) | 29
Completed | 29 | 31 | 28
Not Completed | 1 | 2 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.5mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) | 2.0mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) | 1.5 mg MPA / 0.3 mg CEE (Prempro) | Total
Number analyzed (Participants) | 29 | 32 | 29 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (4.6) | 54.6 (5.6) | 54.1 (4.5) | 55.0 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 32 | 29 | 90
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Black / African American | 3 | 1 | 1 | 5
  White | 9 | 12 | 9 | 30
  Hispanic | 17 | 19 | 19 | 55
Smoking history [Number; unit: participants] — Subjects smoking more than 10 cigarettes per day were excluded from the study.
  participants
    no | 24 | 24 | 25 | 73
    yes | 5 | 8 | 4 | 17
Baseline ambulatory blood pressure [Mean (Standard Deviation); unit: mmHg] — 24-hour mean Ambulatory blood pressure monitoring (ABPM) values at the Baseline visit.
  mmHg
    systolic blood pressure (SBP) | 121.4 (7.6) | 120.9 (10.4) | 122.1 (11.6) | 121.4 (9.9)
    diastolic blood pressure (DBP) | 72.4 (6.7) | 73.1 (7.6) | 73.9 (8.0) | 73.1 (7.4)
Baseline cuff blood pressure [Mean (Standard Deviation); unit: mmHg] — The baseline SBP was to be between 130 and 139 mmHg and DBP ≤ 89 mmHg. The mean SBP values from 2 of the 3 consecutive office cuff measurements during the screening visits were to have been within 12 mmHg and the mean DBP values within 8 mmHg to confirm stability of the blood pressure.
  mmHg
    systolic blood pressure (SBP) | 133.6 (3.2) | 134.3 (2.1) | 133.7 (2.4) | 133.9 (2.6)
    diastolic blood pressure (DBP) | 81.5 (4.7) | 81.7 (4.0) | 80.3 (5.7) | 81.2 (4.8)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] — Height, body weight, and arm circumference were measured at the screening visit and body weight was measured at the screening, treatment phase, and follow-up visits. The same scale was used for all body weight measurements. BMI was measured in kg/m^2.
  Kg/m^2 | 29.1 (5.2) | 27.6 (4.4) | 27.9 (3.4) | 28.2 (4.4)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 8 in Mean 24-hour SBP From the Ambulatory Blood Pressure Monitoring (ABPM) Measurements in Full Analysis Set (FAS) Population
Description: The mean change in 24-hr ambulatory systolic blood pressure (SBP) from Baseline to Week 8 was calculated for the full analysis set. The change from baseline means was adjusted for center and baseline SBP.
Time Frame: Baseline to Week 8
Population: Primary analysis used Full Analysis Set (FAS), which follows ITT principles; no imputation methods used; patients with missing data had no Blood Pressure (BP) values after baseline
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | 0.5mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) | 2.0mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) | 1.5 mg MPA / 0.3 mg CEE (Prempro)
Number analyzed (Participants) | 28 | 32 | 25
mmHg | -1.03 (1.49) | -0.27 (1.35) | 2.18 (1.59)
Statistical Analysis 1: Comparison: 0.5mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) vs 1.5 mg MPA / 0.3 mg CEE (Prempro); Pairwise comparisons among all three treatment groups were performed; both DRSP / E2 group vs MPA /CEE, and the two active doses against each other. Null hypotheses were that there were no differences between groups for each of the three pairwise comparison. Analysis of variance model was used, with terms for treatment, center, and baseline BP values; Test type: Superiority or Other; p = 0.1182, ANCOVA — 0.5 mg DRSP / 1.0 mg E2 vs 1.5 mg MPA / 0.3 mg CEE; No adjustments made for multiple comparisons
Statistical Analysis 2: Comparison: 2.0mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) vs 1.5 mg MPA / 0.3 mg CEE (Prempro); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2224, ANCOVA — 2.0 mg DRSP / 1.0 mg E2 vs 1.5mg MPA / 0.3 mg CEE; No adjustments made for multiple comparisons
Statistical Analysis 3: Comparison: 0.5mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) vs 2.0mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6929, ANCOVA — 0.5 mg DRSP / 1.0 mg E2 vs 2.0 mg DRSP / 1.0 mg E2; No adjustments made for multiple comparisons

2. Primary Outcome: Change From Baseline to Week 8 in Mean 24-hour SBP From the ABPM Measurements in Per Protocol Population
Description: The mean change in 24-hr ambulatory systolic blood pressure (SBP) from Baseline to Week 8 was calculated for the per protocol (PP) population. The change from baseline means was adjusted for center and baseline SBP.
Time Frame: Baseline to Week 8
Population: Primary analysis was Per Protocol Population (PP); no imputation methods used; patients with missing data had no BP values after baseline.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | 0.5mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) | 2.0mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) | 1.5 mg MPA / 0.3 mg CEE (Prempro)
Number analyzed (Participants) | 26 | 28 | 23
mmHg | -1.08 (1.62) | 0.06 (1.50) | 2.82 (1.75)
Statistical Analysis 1: Comparison: 0.5mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) vs 1.5 mg MPA / 0.3 mg CEE (Prempro); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0702, ANCOVA — 0.5 mg DRSP / 1.0 mg E2 vs 1.5 mg MPA / 0.3 mg CEE; No adjustments made for multiple comparisons
Statistical Analysis 2: Comparison: 2.0mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) vs 1.5 mg MPA / 0.3 mg CEE (Prempro); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1980, ANCOVA — 2.0 mg DRSP / 1.0 mg E2 vs 1.5mg MPA / 0.3 mg CEE; No adjustments made for multiple comparisons
Statistical Analysis 3: Comparison: 0.5mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) vs 2.0mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5777, ANCOVA — 0.5 mg DRSP / 1.0 mg E2 vs 2.0 mg DRSP / 1.0 mg E2; No adjustments made for multiple comparisons

3. Secondary Outcome: Change From Baseline to Week 8 in Mean 24-hour DBP From the ABPM Measurements
Description: The mean change in 24-hr Diastolic Blood Pressure (DBP) from Baseline to Week 8 was calculated for the full analysis set.
Time Frame: Baseline to Week 8
Population: Primary analysis used FAS; no imputation methods used; patients with missing data had no BP values after baseline
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | 0.5mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) | 2.0mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) | 1.5 mg MPA / 0.3 mg CEE (Prempro)
Number analyzed (Participants) | 28 | 32 | 25
mmHg | -1.19 (1.02) | -0.91 (0.93) | 0.57 (1.09)

4. Secondary Outcome: Change From Baseline to Week 8 in Office Cuff SBP and DBP at Trough
Description: Seated systolic and diastolic office cuff blood pressures were taken at each visit; the mean of three readings were used at each timepoint.
Time Frame: Baseline to Week 8
Population: Primary analysis used FAS; no imputation methods used; patients with missing data had no BP values after baseline
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | 0.5mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) | 2.0mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) | 1.5 mg MPA / 0.3 mg CEE (Prempro)
Number analyzed (Participants) | 29 | 32 | 28
mmHg
  Systolic Blood Pressure (SBP) | -5.25 (1.54) | -6.02 (1.44) | -4.20 (1.59)
  Diastolic Blood Pressure (DBP) | -1.34 (1.13) | -0.36 (1.05) | 0.33 (1.15)

5. Secondary Outcome: Change From Baseline to Week 8 in Mean Day Time, Mean Nighttime and Mean Trough SBP From the ABPM Measurements
Description: Systolic blood pressure means were calculated during the intervals daytime (6 AM - 10 PM); nighttime (10 PM - 6 AM), and trough (mean of last 5 measurements in the 24-hour cycle)
Time Frame: Baseline to Week 8
Population: Primary analysis used FAS; no imputation methods used; patients with missing data had no BP values after baseline; number of subjects analyzed was 27 in the 0.5mg DRSP group for nighttime values
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | 0.5mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) | 2.0mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) | 1.5 mg MPA / 0.3 mg CEE (Prempro)
Number analyzed (Participants) | 28 | 32 | 25
mmHg
  mean daytime | -2.08 (1.49) | -1.06 (1.35) | 1.53 (1.59)
  mean nighttime | 1.57 (1.99) | 1.64 (1.75) | 3.97 (2.06)
  mean trough | -1.91 (1.99) | -1.48 (1.81) | -1.51 (2.15)

6. Secondary Outcome: Change From Baseline to Week 8 in Mean Day Time, Mean Nighttime and Mean Trough DBP From the ABPM Measurements
Description: Diastolic blood pressure means were calculated during the intervals daytime (6 AM - 10 PM); nighttime (10 PM - 6 AM), and trough (mean of last 5 measurements in the 24-hour cycle)
Time Frame: Baseline to Week 8
Population: as for outcome 5
Measure: Median (Standard Error); unit: mmHg
Arm/Group | 0.5mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) | 2.0mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) | 1.5 mg MPA / 0.3 mg CEE (Prempro)
Number analyzed (Participants) | 28 | 32 | 25
mmHg
  mean daytime | -1.95 (1.03) | -1.56 (0.93) | 0.17 (1.10)
  mean nighttime | 0.20 (1.48) | 0.67 (1.30) | 1.75 (1.54)
  mean trough | -1.04 (1.46) | -1.13 (1.32) | -0.30 (1.57)

7. Secondary Outcome: Number of Subjects Who Are Sodium Sensitive at Baseline and Week 8
Description: Sodium sensitivity was defined as ≥ 10 mmHg drop in mean arterial pressure, calculated from the office cuff BP values from Day 1 to Day 3. The number of subjects shifting from sodium sensitive at Baseline to sodium resistant at Week 8 or sodium resistant at Baseline to sodium sensitive at Week 8 by treatment group was reported.
Time Frame: 8 weeks plus 3 days
Population: FAS subjects from the one site which performed the sodium sensitivity analysis
Measure: Number; unit: participants
Arm/Group | 0.5mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) | 2.0mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) | 1.5 mg MPA / 0.3 mg CEE (Prempro)
Number analyzed (Participants) | 9 | 9 | 10
participants
  Baseline | 4 | 3 | 4
  Week 8 | 1 | 2 | 2

8. Secondary Outcome: Change From Baseline to Week 8 in Mean 24-hours ABPM SBP Values, Baseline Mean > 112 mmHg (Posthoc Analysis)
Description: Mean 24-hour ABPM SBP values were calculated in posthoc subgroup analyses for the following subgroups: Baseline mean 24-hour SBP from ABPM >112 mmHg, >116 mmHg, >120 mmHg, >124 mmHg, and >130 mmHg.
Time Frame: Baseline to Week 8
Population: FAS population, for patients with baseline 24-hour ABPM means > 112 mmHg
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 0.5mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) | 2.0mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) | 1.5 mg MPA / 0.3 mg CEE (Prempro)
Number analyzed (Participants) | 23 | 24 | 19
mmHg | -1.9 (8.2) | -1.9 (9.1) | 1.4 (6.3)

9. Secondary Outcome: Change From Baseline to Week 8 in Mean 24-hours ABPM SBP Values, Baseline Mean > 116 mmHg (Posthoc Analysis)
Description: as for outcome 8
Time Frame: Baseline to Week 8
Population: FAS population, for patients with baseline 24-hour ABPM means > 116 mmHg
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 0.5mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) | 2.0mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) | 1.5 mg MPA / 0.3 mg CEE (Prempro)
Number analyzed (Participants) | 20 | 21 | 17
mmHg | -2.4 (7.9) | -2.2 (9.6) | 2.0 (6.4)

10. Secondary Outcome: Change From Baseline to Week 8 in Mean 24-hours ABPM SBP Values, Baseline Mean > 120 mmHg (Posthoc Analysis)
Description: as for outcome 8
Time Frame: Baseline to Week 8
Population: FAS population, for patients with baseline 24-hour ABPM means > 120 mmHg
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 0.5mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) | 2.0mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) | 1.5 mg MPA / 0.3 mg CEE (Prempro)
Number analyzed (Participants) | 17 | 16 | 14
mmHg | -2.6 (8.1) | -3.7 (9.9) | 1.1 (5.8)

11. Secondary Outcome: Change From Baseline to Week 8 in Mean 24-hours ABPM SBP Values, Baseline Mean > 124 mmHg (Posthoc Analysis)
Description: as for outcome 8
Time Frame: Baseline to Week 8
Population: FAS population, for patients with baseline 24-hour ABPM means > 124 mmHg
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 0.5mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) | 2.0mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) | 1.5 mg MPA / 0.3 mg CEE (Prempro)
Number analyzed (Participants) | 11 | 14 | 14
mmHg | -3.4 (6.9) | -4.4 (10.4) | 1.1 (5.8)

12. Secondary Outcome: Change From Baseline to Week 8 in Mean 24-hours ABPM SBP Values, Baseline Mean > 130 mmHg (Posthoc Analysis)
Description: as for outcome 8
Time Frame: Baseline to Week 8
Population: FAS population, for patients with baseline 24-hour ABPM means > 130 mmHg
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 0.5mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) | 2.0mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) | 1.5 mg MPA / 0.3 mg CEE (Prempro)
Number analyzed (Participants) | 4 | 9 | 6
mmHg | -5.2 (10.1) | -4.0 (12.5) | 1.0 (8.0)

ADVERSE EVENTS:
Arm/Group | 0.5mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) | 2.0mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) | 1.5 mg MPA / 0.3 mg CEE (Prempro)
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/32 | 0/29
Other Adverse Events (participants affected / at risk) | 8/29 | 14/32 | 7/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.5mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) (N=29) | 2.0mg DRSP / 1.0mg E2 (Angeliq, BAY86-4891) (N=32) | 1.5 mg MPA / 0.3 mg CEE (Prempro) (N=29)
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 3 | 1
Fatigue (General disorders) | 0 | 2 | 0
Irritability (General disorders) | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 2
Crying (Psychiatric disorders) | 2 | 0 | 0
Breast tenderness (Reproductive system and breast disorders) | 3 | 5 | 2
Metrorrhagia (Reproductive system and breast disorders) | 1 | 6 | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 4 | 4 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0

LIMITATIONS AND CAVEATS:
Small sample size, as this was a pilot study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
(A). PI will provide copy to Sponsor sixty (60) days. Sponsor will have thirty (30) days to review and provide feedback. (B). If proposed publication presents material adverse effect on Sponsor's confidentiality information, then PI shall delay or prevent such publication. (C) In multi-center trial, the investigative data will be pooled and published as a collaborative effort with consent from all parties including the Sponsor.